CLINICAL TRIAL: NCT04417868
Title: Evolution of Cochleovestibular Schwannomas in the Internal Auditory Canal by Volume Measering With aTeslas MRI 3
Brief Title: Evolution of Cochleovestibular Schwannomas
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7560
Record Dates: First submitted 2020-06-02; First posted 2020-06-05 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Schwannoma
Keywords: schwannoma; cochleovestibular schwannomas; cochleovestibular; intra labyrinthine schwannoma
MeSH Terms: conditions — Neurilemmoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Investigators want to know the natural history of the vestibular schwannomas: increasing, decreasing or stability, by monitoring more than 3 MRIs during a span of more than 2 years. They will obtain 3 groups: the volume increasing schwannomas which will be the most important group, the schwannomas that will be stable and a small group where the schwannomas will decrease.

The secondary purpose is that the investigators want to know the threshold values: a minimum volume under which we are sure that the schwannoma will not increase, a maximum value where it will increase and if its evolution can be correlated to clinical or radiological criteria.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* having a typical vestibular schwannoma diagnosis during the first MRI, having a minimum of 3 internal auditory canal MRIs on the same machine (Signa HDxt, General Electric, Strasbourg, France) ) at the Hôpitaux Universitaires de Strasbourg
* patients consenting to participate

Exclusion Criteria:

* intra-labyrinthical extension
* treatment before the 3 MRIs
* no injection of gadolinium
* atypical diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients having a typical vestibular schwannoma diagnosis during the first MRI, having a minimum of 3 internal auditory canal MRIs on the same machine (Signa HDxt, General Electric, Strasbourg, France) ) at the Hôpitaux Universitaires de Strasbourg
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Presence or absence of intra labyrinthine vestibular nerve tumor using T2 FIESTA | 1 hour after the realization of the MRI

CONTACTS AND LOCATIONS:
Locations (1):
- Service Imagerie 1, Srtrasbourg, Strasbourg, France